CLINICAL TRIAL: NCT06546761
Title: Selective Coronary Revascularization in Carotid Artery Disease Patients After Carotid Revascularization (SCORECAD Trial)
Status: Recruiting | Type: Observational
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Latvia RCT/CAD/25062024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Carotid Stenosis; Coronary Artery Disease
MeSH Terms: conditions — Carotid Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assigned to Best Medical Therapy (BMT) alone: Patients who have undergone successful carotid artery revascularization (endarterectomy of stenting) and are assigned to BMT alone within 14 days following revascularization.
- Assigned to Best Medical Therapy (BMT) + coronary CT angiography + CT-FFRct analysis: Patients who have undergone successful carotid artery revascularization (endarterectomy of stenting) and are assigned to BMT plus coronary CT angiography (which must be completed within 14 days of randomization) and FFRct analysis to determine the functional significance of coronary lesions identified on the CT scan.
  Interventions: Diagnostic Test: Coronary CT angiography and FFRct analysis

INTERVENTIONS:
Diagnostic Test: Coronary CT angiography and FFRct analysis — A new non-invasive cardiac diagnostic test, coronary CT-derived fractional flow reserve (FFRCT) provides a unified anatomic and functional assessment of coronary artery disease which can reliably identify ischemia-producing coronary lesions. FFRCT accurately reflects invasively measured FFR and can help guide patient management and coronary revascularization decisions.
  Groups: Assigned to Best Medical Therapy (BMT) + coronary CT angiography + CT-FFRct analysis

SUMMARY:
The primary objective of this study is to determine whether among symptomatic and asymptomatic carotid artery stenosis (CAS) patients with no known coronary artery disease (CAD) who had undergone carotid artery revascularization (endarterectomy of stenting) a strategy of best medical therapy (BMT) plus selective coronary revascularization based on FFRct assessment of lesion-specific coronary ischemia can reduce adverse cardiac events and improve survival compared to BMT alone. Lesion-specific coronary ischemia is defined as FFRCT ≤0.80 distal to stenosis in a major (≥2 mm) coronary artery with severe ischemia defined as FFRCT ≤0.75.

DETAILED DESCRIPTION:
This study targets a population of patients with symptomatic or asymptomatic carotid artery stenosis (CAS) (symptomatic to asymptomatic in 1:1 ratio) and no prior cardiac history, no myocardial infarction, no coronary angiography or coronary computed tomography angiography (CTA), and no coronary revascularization (PCI or CABG) who have undergone successful carotid artery revascularization with planned post-operative best medical therapy. Within 14 days following carotid revascularization, patients will be randomly assigned to BMT alone or BMT plus coronary CT angiography (which must be completed within 14 days of randomization) and FFRct analysis to determine the functional significance of coronary lesions identified on the CT scan. Results of the CT scan and FFRCT analysis in patients randomized to the CT-FFRct group, will be provided to treating physicians to help guide patient management with Vascular Heart Team consideration for coronary angiography and revascularization as appropriate for each patient. Coronary revascularization (PCI or CABG), if indicated, is strongly recommended within 3 months from the randomization. Clinical follow up (based on date of randomization) is planned 6 months, one and 2 years. Additional long-term follow up out to 5-years is planned for participating centers. An independent academic clinical events committee will adjudicate all endpoints in a blinded manner. The definition of outcome events will be in accordance with Academic Research Consortium-2 consensus document.

ELIGIBILITY:
Inclusion Criteria:

1. Inform consent obtained before any study-related activities;
2. Age above or equal to 50 years with symptomatic or asymptomatic critical carotid stenosis (symptomatic patients with at least Rankin III) which has been successfully revascularized by carotid endarterectomy or stenting within the past 14 days;
3. Willing and able to undergo coronary CTA scan within 14 days of randomization and agrees to submission of CTA data set for HeartFlow FFRct analysis with results made available to treating physician.

Exclusion Criteria:

1. Known CAD, history of MI, prior coronary revascularization (PCI or CABG);
2. Patient underwent coronary angiography or coronary CTA before the randomization;
3. Known history of 2nd or 3rd degree heart block; sick sinus syndrome; long QT syndrome;
4. History of severe asthma, severe or bronchodilator-dependent Chronic obstructive pulmonary disease (COPD);
5. Severe congestive heart failure (NYHA III or IV);
6. Severe arrhythmia, prior pacemaker or internal defibrillator lead implantation;
7. Impaired chronic renal function (EPI-GFR<30ml/min);
8. Subjects with known anaphylactic allergy to iodinated contrast;
9. Pregnancy or unknown pregnancy status in subject of childbearing potential;
10. Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, or acute pulmonary edema;
11. Any active, serious, life-threatening disease with a life expectancy of less than 2 years;
12. Any active infection;
13. Inability to comply with study procedures;
14. Contraindication for guideline-guided long-term antiplatelet/anticoagulation regime after PCI/CABG;
15. Large neurologic deficit (Rankin scale >III);
16. Participation in any interventional clinical study within 30 days prior to screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic or asymptomatic carotid artery stenosis (CAS) (symptomatic to asymptomatic in 1:1 ratio) and no prior cardiac history, no myocardial infarction, no coronary angiography or coronary CTA, and no coronary revascularization (PCI or CABG) who have undergone successful carotid artery revascularization with planned post-operative best medical therapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2029-06-25 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 2 years
  A composite of cardiac death, myocardial infarction (MI) or urgent coronary revascularization

SECONDARY OUTCOMES:
Major Adverse Cardiac Events and survival | 2 years
  Cardiac death, cardiovascular death, myocardial infarction (MI), urgent coronary revascularization, all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT06546761/Prot_000.pdf